CLINICAL TRIAL: NCT00003840
Title: A Phase I Study of DTGM Fusion Protein (IND BB#8153) in Relapsed and Refractory Adult Acute Myeloid Leukemia (AML)
Brief Title: DTGM Fusion Protein in Treating Patients With Recurrent or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CCCWFU-22300; CDR0000066998 (Registry Identifier: PDQ (Physician Data Query)); CCCWFU-22198; NCI-H99-0027
Record Dates: First submitted 1999-11-01; First posted 2004-04-12 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute

INTERVENTIONS:
Biological: DTGM fusion protein

SUMMARY:
RATIONALE: DTGM fusion protein may be able to locate cancer cells and stop them from growing.

PURPOSE: Phase I/II trial to study the effectiveness of DTGM fusion protein in treating patients who have recurrent or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of DTGM fusion protein in patients with recurrent or refractory adult acute myeloid leukemia. II. Determine the dose-limiting toxic effects of this regimen in these patients. III. Measure the pharmacokinetics of this regimen in these patients. IV. Evaluate the response rate at the maximum tolerated dose and immune responses in patients treated with this regimen. V. Correlate in vitro sensitivity of leukemic blasts to this regimen with the response rate in these patients. VI. Correlate tumor necrosis factor genetic polymorphisms with toxicity profiles and dose-limiting toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to serum level of anti-DTGM antibody titer (2 mg/L or less vs greater than 2 mg/L). Patients receive DTGM fusion protein IV over 15 minutes on days 1-5. Patients with a partial response are eligible for retreatment. Cohorts of 3-6 patients receive escalating doses of DTGM fusion protein until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with DTGM fusion protein at the MTD. Patients are followed monthly until disease progression.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically, morphologically, or cell surface marker confirmed adult acute myeloid leukemia (AML) Recurrent or refractory after at least 1 prior induction therapy OR Relapsed after remission of less than 1 year duration Antecedent myelodysplasia that has evolved to AML allowed Ineligible for allogeneic stem cell transplantation or failed prior transplantation No CNS leukemia

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC no greater than 10,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases less than 5 times upper limit of normal Albumin at least 3 g/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: Cardiac ejection fraction at least 50% normal No myocardial infarction within the past 6 months No disseminated intravascular coagulation Pulmonary: FEV1 at least 70% normal Other: No uncontrolled infections No other concurrent serious medical problems or psychiatric disorders No prior severe penicillin allergy (hives or anaphylactic reactions) Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No concurrent growth factors Chemotherapy: See Disease Characteristics Recovered from prior chemotherapy Prior hydroxyurea or low-dose cytarabine (less than 100 mg subcutaneously) to lower blast counts allowed if discontinued on day 1 of study therapy No concurrent antineoplastic chemotherapy Endocrine therapy: Concurrent corticosteroids allowed, including antiemetics Radiotherapy: Recovered from prior radiotherapy No concurrent radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2002-09 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur E. Frankel, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States